CLINICAL TRIAL: NCT03039881
Title: Blinded Observational Study to Evaluate a Non-Invasive Respiratory Volume Monitor in the Post-Anesthesia Care Unit and on the General Hospital Floor
Brief Title: Evaluation of Non-Invasive Respiratory Volume Monitor
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Collaborators: Respiratory Motion, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 11544
Record Dates: First submitted 2017-01-27; First posted 2017-02-01 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Monitoring for Low Minute Ventilation Post Surgery
Keywords: Minute ventilation, ExSpiron monitor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Device: Yes

INTERVENTIONS:
Device: Non-Invasive Respiratory Volume Monitor — The device requires the application of a monitoring PadSets to the patient's skin similar to EKG electrodes and, as such, poses minimal risk.

SUMMARY:
This observational study investigates the validity and utility of a new, non-significant risk, FDA approved respiratory monitor, ExSpiron, in the perioperative course of patients undergoing elective surgery under general anesthesia. The study patients will be monitored before, during and after surgery, in post-anaesthesia care unit (PACU) and recovery room for the first post-operative night. The physiologic data will not be used or influence the standard of care for subjects. It is anticipated that this monitor may be able to improve perioperative care in the future.

DETAILED DESCRIPTION:
Aim and Hypotheses Currently, there is no objective measure of early respiratory indicators for developing respiratory compromise in surgical patients. Current respiratory assessment in non-intubated patients relies on oximetry data and subjective clinical assessment. Pulse oximetry has been extremely helpful in recognizing oxygen desaturations but it is a late indicator of respiratory decline. New advances in technology and digital signal processing have led to the development of an impedance based Respiratory Volume Monitor (RVM). The RVM (ExSpiron™, Respiratory Motion, Inc.; Waltham, MA) has been shown to provide accurate real-time, continuous, non-invasive measurements of tidal volume (TV), minute ventilation (MV) and respiratory rate (RR) in general patient population.

Hypotheses

Primary:

Low minute ventilation (LMV) defined as sustained LMV<40% minute ventilation predicted (MVPRED) based on IBW following opioid administration correlates with adverse clinical outcomes in PACU or on the floor including:

* O2 desaturation, atelectasis, respiratory status requiring advanced monitoring
* respiratory interventions such as O2 administration, continuous positive airway pressure CPAP, BiPAP,
* incidence of ICU transfer and/or increase in PACU and/or general hospital floor (GHF) length of stay (LOS).

Secondary:

* 1. Decreased MV defined as sustained MV<80% MVPRED based on IBW before opioid administration correlates with adverse clinical outcomes as defined above.
* 2. Patients with decreased MV prior to opioid administration will be more likely to develop LMV after standard opioid administration compared to patients with normal MV defined as MV ≥ 81% MVPRED based on ideal body weight (IBW)

Rationale Continuous respiratory monitoring using the ExSpiron System will be particularly beneficial to patients in the post-anesthesia environment. Assessment and management of respiratory function and early intervention when indicated is a multifaceted, complex task often complicated by the lack of a cohesive and continuous monitoring system to guide clinical decisions. The ExSpiron system is designed for these patients and is intended to address some of the limitations of the current generation of hospital monitors and to provide healthcare providers with continuous real-time data regarding the patient's respiratory status. Recent data has shown that stratification of patients based on the RVM's MV as % of predicted MV (MVPRED), prior to opioid dosing has made it possible to identify patients who are at risk for further decreases in MV and opioid-induced respiratory depression (OIRD).

1. In the spontaneously breathing, non-ventilated patient, current monitoring devices do not provide continuous, objective non-invasive, continuous real time information of the important respiratory parameters TV, MV & RR.
2. Current monitoring of non-intubated patients mostly relies on subjective clinical assessment, oximetry data, and rarely end-tidal carbon dioxide CO2 measurements. In appropriate clinical settings, the ExSpiron system can provide direct quantitative measure of ventilation parameters for use in clinical assessment and trend prediction as well as response to medications and other interventions to allow for more efficient clinical decision making.
3. Current technologies do not provide for a continuity of care between the PACU and the general hospital floor.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing surgery with general anesthesia and positive pressure ventilation, patient's ≥80 pounds and who are able to give informed consent.

Exclusion Criteria:

* Patients unable to give informed consent. Any patient whose condition or procedure will not allow for placement of the electrode PadSet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective surgery with general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-01-09 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Low minute ventilation | Post-operatively in PACU and general patient' floor up to 24 hours after completion of surgery
  Low minute ventilation (LMV) defined as sustained LMV<40% minute ventilation predicted (MVPRED) based on IBW following opioid administration correlates with adverse clinical outcomes in PACU and on the floor

CONTACTS AND LOCATIONS:
Overall Officials: Iwona Bonney, PhD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No